CLINICAL TRIAL: NCT02759497
Title: Evaluation of Serum Amyloid A in Early Diagnosis of Spontaneous Bacterial Peritonitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sherief Abd-Elsalam, Consultant liver and GIT diseases- Tanta university hospital, Tanta University
Other Study IDs: sbp diagnosis
Record Dates: First submitted 2016-05-01; First posted 2016-05-03 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Spontaneous Bacterial Peritonitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Serum amyloid A level in SBP: serum amyloid A level
  Interventions: Other: serum amyloid A level
- Serum amyloid A level in cirrhosis: Serum amyloid A level
  Interventions: Other: serum amyloid A level

INTERVENTIONS:
Other: serum amyloid A level — serum amyloid A level (SAA)

SUMMARY:
One of the most common and serious complications in decompensated cirrhotic patients (DCPs) is bacterial infection.The most common infections in DCPs are cases of spontaneous bacterial peritonitis (SBP), which account for 40% 70% of cases, followed by urinary tract infections, pneumonia and cellulitis.

Serum amyloid A (SAA) and C-reactive protein (CRP) are acute-phase proteins predominantly produced and secreted by hepatocytes. Other cells including lymphocytes, monocytes, and macrophages can also produce these proteins. The induction of SAA and CRP synthesis is triggered by a number of cytokines, chiefly IL-6, which is released from a variety of cell types, but mainly from macrophages and monocytes at inflammatory sites

DETAILED DESCRIPTION:
Increased serum CRP and SAA levels have been found in a number of disorders, including bacterial infections, malignancies tissue injuries and tissue rejection. Therefore, new studies of early diagnosis, prevention and treatment are needed to improve clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* • Decompansated cirrhosis with ascites, defined by a combination of any of the following:

  * Laboratory findings
  * Endoscopic results
  * Ultrasound
  * Histology

Exclusion Criteria:

* Creatinine>1.5 mg/dl
* Other infection e.grespiratory,UTI ,gastrointestinal and skin infection.
* Hepatocellular carcinoma
* Other extrahepatic malignancy e.g ; chest
* Any significant psychiatric illness or other medical comorbidity.
* Any degenerative diseases.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Decompensated cirrhosis with SBP Decompensated cirrhosis without SBP
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-03; Primary Completion 2020-10 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Number of patients with elevated serum amyloid A | 6months

CONTACTS AND LOCATIONS:
Overall Officials: Rehab Badawi, Consultant, Principal Investigator — Hepatology and gastroenterology dept.-Tanta; Sherief Abd-Elsalam, Consultant, Study Chair — Division of Gastroenterology and Hepatology- Tanta; Walaa Elkhalawany, Consultant, Study Chair — Hepatology and gastroenterology dept.-Tanta; Reham Elkhouly, Consultant, Study Chair — Hepatology and gastroenterology dept.-Tanta; Mona Watany, Consultant, Study Chair — clinical pathology dept.-Tanta; Samah Soliman, Consultant, Study Chair — Hepatology and gastroenterology dept.-Tanta; Mai Khalaf, resident, Study Chair — hepatology dept.-Tanta
Locations (1):
- Sherief Abd-Elsalam, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided